CLINICAL TRIAL: NCT05426850
Title: Circulating Tumor DNA-based Minimal Residual Disease (MRD) Assessment in Local Advanced Esophageal Squamous Cell Carcinoma Treated by Definitive Concurrent Chemoradiotherapy
Brief Title: ctDNA-based MRD Assessment in Local Advanced Esophageal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Other Study IDs: ESO-Shanghai16
Record Dates: First submitted 2022-05-24; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ctDNA(+) Cohort: ctDNA(+) Cohort in pretreatment and posttreatment plasma samples was defined by accessing the presence of one or more mutations identified in match tumor samples.
- ctDNA(-) Cohort: ctDNA(-) Cohort in pretreatment and posttreatment plasma samples was defined by the absence of one or more mutations identified in match tumor samples.

SUMMARY:
To analyze the relationship between the dynamic changes of circulating tumor DNA (ctDNA) and tumor relapse of esophageal squamous cell carcinoma treated by concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old.
2. ECOG 0-1.
3. Esophageal squamous cell carcinoma confirmed by pathology.
4. No radiotherapy, chemotherapy, or other treatments prior to enrollment.
5. Locally advanced esophageal squamous cell carcinoma (II-IVa, IVB with supraclavicular lymph node metastasis).
6. No severe abnormal hematopoietic, cardiac, pulmonary, renal, hepatic function, or immunodeficiency.
7. Informed consent signed.

Exclusion Criteria:

1. Less than 50.4Gy/28fx of radiotherapy dose.
2. Without Concurrent chemotherapy.
3. Pregnant or breastfeeding women or fertile patients who refused to use contraceptives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local advanced esophageal squamous cell carcinoma treated by definitive concurrent chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between ctDNA status after chemoradiotherapy and relapse. | ctDNA will be tested within 1 year after chemoradiotherapy
  To assess if recurrent esophageal cancer is detectable earlier by ctDNA positive in plasma.

SECONDARY OUTCOMES:
Changes of ctDNA status. | before and at the end of radiotherapy (+1 week); at the end of consolidation chemotherapy (+1 week); at 2 weeks, 1 month, 3 months, 6 months, 9 months, 1 year after dCCRT.
  To dynamically evaluate the ctDNA status at baseline, during treatment and follow-up.
Overall survival (OS). | through study completion, an average of 2 years.
  To compare OS in ctDNA(+) patients and ctDNA(-) patients.
Relapse-free survival (RFS) and progression-free survival (PFS). | through study completion, an average of 2 years.
  To compare RFS and PFS in ctDNA(+) patients and ctDNA(-) patients.
Relationships between radiomics features, ctDNA status and relapse. | through study completion, an average of 2 years.
  To assess if recurrent esophageal cancer is detectable earlier by ctDNA positive in plasma compared to traditional radiographic methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai cancer center, Shanghai, Shanghai Municipality, China